CLINICAL TRIAL: NCT03522129
Title: A Pilot Study to Evaluate the Effect of CT1812 Treatment on Amyloid Beta Oligomer Displacement Into CSF in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Study to Evaluate the Effect of CT1812 Treatment on Amyloid Beta Oligomer Displacement Into CSF in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG0104
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Phase 1b, randomized, double-blind, placebo-controlled parallel-group trial in adults with mild to moderate AD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind for study site and participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Treatment- CT1812 560 mg (Active Comparator)
  Interventions: Drug: CT1812
- Active Treatment- CT1812 280 mg (Active Comparator)
  Interventions: Drug: CT1812
- Active Treatment- CT1812 90 mg (Active Comparator)
  Interventions: Drug: CT1812
- Placebo Comparator - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT1812 — Active Study Drug
  Other Names: Study Drug
  Arms: Active Treatment- CT1812 280 mg; Active Treatment- CT1812 560 mg; Active Treatment- CT1812 90 mg
Drug: Placebo — Non-active study drug
  Other Names: Matching Placebo
  Arms: Placebo Comparator - Placebo

SUMMARY:
This is a multi-center, Phase 1b, randomized, double-blind, placebo-controlled parallel-group trial in adults with mild to moderate AD.

DETAILED DESCRIPTION:
This is a multi-center, Phase 1b, randomized, double-blind, placebo-controlled parallel-group trial in adults with mild to moderate AD. The primary endpoint is the change from the baseline CSF Amyloid beta oligomer concentration after dosing with CT1812 versus placebo. The change from baseline will be measured through a number of exploratory endpoints as indicated below. For each subject, the baseline CSF oligomer concentration will be computed as the average of the measurements from hours -4, -3, -2 and -1 and 0.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects may be included in the study only if they meet all of the following criteria:

1. Men, and women of non-childbearing potential, 50-85 years of age inclusively, with a diagnosis of mild to moderate Probable Alzheimer's Disease Dementia according to the 2011 NIA-AA criteria and at least a 6 month decline in cognitive function documented in the medical record.

   1. a. Non-childbearing potential for women is defined as postmenopausal [last natural menses greater than 24 months; in women under age 55, menopausal status will be documented with serum follicle stimulating hormone (FSH) test] or undergone a documented bilateral tubal ligation or hysterectomy
   2. b. Male participants who are sexually active with a woman of childbearing potential must agree to use condoms during the trial unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of: intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap.
2. Neuromaging (MRI) obtained during screening consistent with the clinical diagnosis of Alzheimer's disease and without findings of significant exclusionary abnormalities (see exclusion criteria, number 3).
3. MMSE 18-26 inclusive. Subjects must, in the opinion of the investigator, be able to comply with study procedures and must understand the consent process. The investigator will use his or her clinical judgment in conjunction with the cognitive screening assessments to determine whether the subject meets these criteria in a manner that is consistent with local clinical practice and standards. Subjects with borderline low MMSE at screening may undergo repeat MMSE administration if extenuating circumstances were present at original assessment.
4. A positive amyloid scan (florbetaben F18, florbetapir F18, or flutametamol F18) at screening or within prior 12 months, as read by the certified, site-designated PET scan reader.
5. Must consent to apolipoprotein E (ApoE) genotyping.
6. Subjects must have a caregiver or study partner who can participate in all clinic visits.
7. Patients living at home or in the community (assisted living acceptable).
8. Able to swallow CT1812 capsules.
9. Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening.
10. Subjects must be capable of providing either written informed consent to the study procedures and for use of protected health information [Health Insurance Portability and Accountability Act (HIPAA) Authorization, if applicable]. Written informed consent also shall be obtained from the responsible caregiver or study partner. All consent processes must be undertaken in the presence of a witness and prior to any study procedures.
11. Subjects shall be generally healthy with mobility (ambulatory or ambulatory-aided, i.e., walker or cane), vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures.
12. Must be able to complete all screening evaluations.

EXCLUSION CRITERIA:

Subjects will be excluded from the study if any of the following conditions apply:

1. Hospitalization or change of chronic concomitant medication within one month prior to screening.
2. Patients living in a continuous care nursing facility
3. Screening MRI of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor such as meningioma). If a small incidental meningioma is observed, the medical monitor may be contacted to discuss eligibility.
4. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Jacob-Creutzfeld Disease, Down syndrome, etc.);
   2. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.);
   3. Seizure disorder; or
   4. Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism.) Present vitamin B12 or folate deficiency or other laboratory abnormalities of possible clinical significance should be discussed with medical monitor to determine eligibility.
5. A current DSM-V diagnosis that would interfere with the subject's ability to participate in the study. Patients with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
6. Any prior history of suicidal thoughts or behavior that are believed by the investigator to represent a current safety risk.
7. Clinically significant, advanced or unstable disease that may interfere with outcome evaluations, such as:

   1. Chronic liver disease, liver function test abnormalities or other signs of hepatic insufficiency (ALT, AST, > 1.5 ULN);
   2. Respiratory insufficiency;
   3. Renal insufficiency, defined as eGFR <40 mL/min based on the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula, https://www.mdcalc.com/ckd-epi-equations-glomerular-filtration-rate-gfr Heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within six months before screening). If a subject has a history of heart disease of questionable clinical significance, the medical monitor may be contacted to discuss eligibility.
   4. Bradycardia (<50 beats/min.) or tachycardia (>100 beats/min.). Otherwise healthy subjects with borderline bradycardia may be discussed with the medical monitor to determine eligibility.
   5. Poorly managed hypertension (systolic >160 mm Hg and/or diastolic >95 mm Hg) or hypotension (systolic <90 mm Hg and/or diastolic <60 mm Hg); or
   6. Uncontrolled diabetes defined by HbA1c >7.5
8. History of cancer within 3 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months.
9. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for Hepatitis B surface antigen [HbsAg] or anti-Hepatitis C [HCV] antibody).
10. Clinically significant abnormalities in screening laboratory tests, including:

    1. hematocrit less than 35% for males and less than 32% for females
    2. platelet cell count of < 120,000/uL,
    3. INR >1.4 or other coagulopathy, confirmed by repeat analysis, or
    4. lymphocyte count less than 1200/ul
11. Disability that may prevent the patient from completing all study requirements (e.g. blindness, deafness, severe language difficulty, etc.).
12. Within 4 weeks of screening visit or during the course of the study, concurrent treatment with antipsychotic agents, antiepileptics, centrally active anti-hypertensive drugs (e.g., clonidine, l-methyl dopa, guanidine, guanfacine, etc.), sedatives, opioids, mood stabilizers (e.g., valproate, lithium); or benzodiazepines, with the following exceptions:

    1. benzodiazepines must not be administered within 5 half-lives of cognitive testing;
    2. administration of selective serotonin re-uptake inhibitors (SSRI) may be continued if doses have been stable for 60 days prior to Screening;
    3. low dose lorazepam may be used for sedation prior to MRI scan for those patients requiring sedation. At the discretion of the investigator, 0.5 to 1 mg may be given orally prior to scan with a single repeat dose given if the first dose is ineffective. No more than a total of 2 mg lorazepam may be used for the MRI scan.
13. Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. small bowel disease, Crohn's disease, celiac disease, or liver disease.)
14. Nootropic drugs except for AD meds (acetylcholinesterase inhibitors and memantine) stable for at least 30 days
15. Suspected or known drug or alcohol abuse, i.e. more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day indicated by elevated MCV significantly above normal value at screening.
16. Suspected or known allergy to any components of the study treatments.
17. Enrollment in another investigational study or intake of investigational drug within the previous 30 days or five half lives of the investigational drug, whichever is longer.
18. Intake of drugs or substances potentially involved in clinically significant inhibition or induction of CYP3A4 or P-gp mediated drug interactions with CT1812, within 4 weeks or five half-lives of the interacting drug prior to administration of CT1812 and throughout the course of the study. Grapefruit juice should be avoided in the two weeks prior to dosing. See Appendix A and Appendix B for a complete list of prohibited substances.
19. Previous exposure to anti Aβ vaccines.
20. Exposure to passive immunotherapies for AD (e.g. monoclonal antibodies) within the previous 180 days to dosing, or BACE inhibitors within the previous 30 days to dosing..
21. Contraindication to undergoing an LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; international normalized ratio (INR) > 1.4 or other coagulopathy; platelet count of <120,000/μL; infection at the desired lumbar puncture site; taking anti-coagulant medication within 90 days of screening (Note: low dose aspirin is permitted); degenerative arthritis of the lumbar spine; suspected non-communicating hydrocephalus or intracranial mass; prior history of spinal mass or trauma.
22. Positive assay for Lyme disease if a screening lumbar puncture is conducted and includes this measurement.
23. Any condition, which in the opinion of the investigator or the sponsor makes the patient unsuitable for inclusion.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Measuring the displacement of Amyloid beta oligomers into cerebrospinal fluid (CSF) | 48 hours
  evidence of oligomer displacement as demonstrated by a clear rise in CSF oligomer concentration relative to baseline and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Galley, Study Director — Cognition Therapeutics, Inc.
Locations (2):
- United States (2):
  - Clinilabs Drug Development Corporation, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] LaBarbera KM, Sheline YI, Izzo NJ, Yuede CM, Waybright L, Yurko R, Edwards HM, Gardiner WD, Blennow K, Zetterberg H, Borjesson-Hanson A, Morgan R, Davis CS, Guttendorf RJ, Schneider LS, DeKosky S, LeVine H 3rd, Grundman M, Caggiano AO, Cirrito JR, Catalano SM, Hamby ME. A phase 1b randomized clinical trial of CT1812 to measure Abeta oligomer displacement in Alzheimer's disease using an indwelling CSF catheter. Transl Neurodegener. 2023 May 12;12(1):24. doi: 10.1186/s40035-023-00358-w. No abstract available. PMID 37173791